CLINICAL TRIAL: NCT05194306
Title: Evaluation of the Safety and Performance of Perla® Preservation Solution for Donor Liver and Kidney for Transplantation
Brief Title: PERTRIAL - Perla® Preservation Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Life Solutions (Industry)
Collaborators: Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP001A
Record Dates: First submitted 2021-12-14; First posted 2022-01-18 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-01

CONDITIONS: Organ Transplant; Ischemic Reperfusion Injury
Keywords: Cold Preservation Solution; Ischemic Reperfusion Injury; Organ Transplant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perla® Cold Preservation solution (Experimental): Perla® is a Cold Preservation Solution, with purpose to wash out, preserve during transport liver and kidney grafts in optimal conditions from the donor to the recipient.
  Interventions: Drug: Perla® Cold Preservation solution

INTERVENTIONS:
Drug: Perla® Cold Preservation solution — Perla® must be cooled to 2° to 6 °C prior to use. The cold Preservation Solution is used to flush the isolated organ immediately before removal from the donor and/or immediately after removal from the donor. The solution is then left in the organ vasculature during hypothermic storage and transportation.

SUMMARY:
Perla® is a Cold Preservation Solution, with purpose to wash out, preserve during transport liver and kidney grafts in optimal conditions from the donor to the recipient.

The purpose of the PERTRIAL clinical investigation is to demonstrate the Performance and Safety of Perla® Cold Preservation solution.

ELIGIBILITY:
Donor kidney / liver eligibility criteria:

Inclusion Criteria:

* Donor kidney / liver suitable for preservation
* Donor age equal or over 18 years old
* Donor meets one of the following conditions:
* Donor after brain death (DBD), standard and extended criteria (SCD & ECD)
* Donor after circulatory death (DCD), cardiac arrest Maastricht classification III (awaiting cardiac arrest, controlled)

Exclusion Criteria:

* Donor participating at the same time in another Clinical Investigation

Recipient eligibility criteria:

Inclusion Criteria:

* Patient registered primary kidney or liver transplant candidate, male or female
* Patient ages ≥ 18 years old
* Patient who has signed written informed consent

Exclusion criteria:

Patient recipient will not be included if any of the following conditions exists:

* Prior solid organ or bone marrow transplant
* Multi-organ transplant
* Contraindications to transplantation (Active infection, active malignancy, pregnant females, females intending to get pregnant, or not willing to use a secure contraceptive method)
* Participation in another clinical trial
* Patient unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-12-11 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Graft Function Rate (Kidney & Liver) | 7 days post transplant

SECONDARY OUTCOMES:
Graft survival (Kidney & Liver) | 7 days post-transplant
Graft survival (Kidney & Liver) | 14 & 30 days post-transplant
Rate of an event or serious adverse device effects (Kidney & Liver) | within 30 days post-transplant
Evaluation of patient anxiety (Kidney & Liver) | pre-transplant
  The patient will complete the HAD scale ("Hospital Anxiety and Depression Scale") after signing his/her consent before the transplant.
Duration of delayed graft function (Kidney) | within 30 days post-transplant
Rate of functional delayed graft function (f-DGF) (Kidney) | within 7 days post-transplant
Daily serum creatinine (Kidney) | 7 days post-transplant, or until the patient is discharged - whichever is earliest
Peak level of serum AST (Liver) | within 7 days post-transplant
Post-reperfusion syndrome (Liver) | during operative procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalario Universitario A Coruña (CHUAC), A Coruña, Spain